CLINICAL TRIAL: NCT00873652
Title: An Observational Study of Children Immunised in Infancy Against Hepatitis B Virus, Evaluating the Persistence of Immunity and the Immune Response to a Scheduled Booster Dose of Hepatitis B Vaccine
Brief Title: Observational Study of Immune Response to Hepatitis B Childhood Booster
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OVG 2008/5
Record Dates: First submitted 2009-01-27; First posted 2009-04-01 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: Hepatitis B vaccine; Booster dose; Persistence; Immune response; Healthy children
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B; Hepatitis B Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Engerix B®, a recombinant hepatitis B vaccine — Single 0.5 ml dose intramuscularly into the deltoid muscle
  Other Names: Hepatitis B Vaccine (Recombinant)

SUMMARY:
The UK immunisation guidelines recommend that children immunised with an accelerated course of hepatitis B vaccine (i.e. vaccination at 0, 1, 2 and 12 months) receive an additional booster dose of vaccine in later childhood (usually at 3 1/2 years of age). The primary objective of this study is to to assess what proportion of these children have 'protective' concentrations (10mIU/ml) of hepatitis B specific antibodies before and after the booster dose of hepatitis B vaccine.

DETAILED DESCRIPTION:
This is an observational, open label study of children immunised in infancy against Hepatitis B virus (HBV),evaluating the persistence of immunity and the immune response to a scheduled booster dose of Hepatitis B vaccine.

Children eligible/overdue for their pre school HBV vaccine booster will be identified by reviewing clinical records at the John Radcliffe Hospital. The parents/legal guardians of these children will be written to and advised that their child should receive/ have received a booster dose of HBV vaccine. This letter will also inform parents/ legal guardians that they have the option of participating in this study looking at the persistence of HBV vaccine induced antibodies through early childhood and the response to a booster dose of HBV vaccine, and that this study will be conducted by the Oxford Vaccine Group in the participants' homes. Parents will be advised that if they do not wish to take part in this research study they should arrange to contact their GP to discuss whether their child requires a booster dose of hepatitis B vaccine.

For participants the study will consist of two visits at a four week interval(visit 1 and visit 2). If the parents/guardians then sign the consent form a medical and immunisation history will be taken and a medical examination will be undertaken if indicated. If no exclusion criteria are identified, the child will be enrolled in the study. A 6ml blood sample will be taken from the child and single booster dose of Hepatitis B vaccine will be administered.

For all children receiving the booster dose of vaccine and their GP, practice nurse and child health department will be informed. If the child is also due for their other pre-school booster vaccines (the 4 in 1 Diphtheria, tetanus, tetanus and polio vaccine, the combined Hib-MenC vaccine and the combined measles, mumps, rubella vaccine (MMR)) these will also be offered, but will not form part of the study assessment.

At the second visit following a confirmation of ongoing consent for the study the first eligibility for inclusion will be checked along with the occurrence of any serious adverse events, 6mls of blood will be drawn from the participant.

Blood samples will be used for antibody analysis by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian is willing and able to give informed consent for participation in the study.
* Male or Female, aged 3 years 4 months or above.
* Commenced Hepatitis B post exposure prophylaxis at birth.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Parent/guardian is not willing or able to give informed consent for participation in the study.
* The child is currently enrolled in any other interventional research study
* History of a confirmed anaphylactic reaction to a previous dose of hepatitis B containing vaccine or a confirmed reaction to any component of the vaccine
* Evidence of infection with HBV on previous blood tests.
* Previous receipt of booster doses of HBV vaccine within the 2 years prior to study enrolment.
* Significant renal or hepatic impairment.
* Participant who is terminally ill.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the patient/participant at risk because of participation in the study, or may influence the result of the study, or the patient/participant's ability to participate in the study.

Ages: 41 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children have been recorded as having commenced an accelerated course of HBV vaccine between the years 2000 and 2006
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The percentage of participants completing an accelerated course of hepatitis B vaccination with 10 IU/ml Hepatitis B surface antigen specific antibodies (antiHBs) before and after the 'pre-school' booster dose of Hepatitis B vaccine. | immediately prior to vaccination and 4 weeks post vaccination

SECONDARY OUTCOMES:
To evaluate the percentage of participants who had serum antiHBs concentrations < 10 IU/ml at visit 1 who had a rise in serum antiHBs to 10 IU/ml at visit 2. | immediately prior to vaccination and 4 weeks post-vaccination
To evaluate the percentage of participants who had serum antiHBs concentrations < 10 IU/ml at visit 1 who had a rise in serum antiHBs to 100 IU/ml at visit 2. | immediately prior to vaccination and 4 weeks post-vaccination
To evaluate the serum antiHBs geometric mean concentrations (GMCs) at visit 1 and visit 2. | immediately prior to vaccination and 4 weeks post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Snape, MBBS, FRCPCH, Principal Investigator — Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford OX3 7LJ
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Yates TA, Paranthaman K, Yu LM, Davis E, Lang S, Hackett SJ, Welch SB, Pollard AJ, Snape MD. UK vaccination schedule: persistence of immunity to hepatitis B in children vaccinated after perinatal exposure. Arch Dis Child. 2013 Jun;98(6):429-33. doi: 10.1136/archdischild-2012-302153. Epub 2013 Mar 9. PMID 23476003